CLINICAL TRIAL: NCT00937807
Title: Hemodynamic Stability During Carotid Endarterectomy Under General Anesthesia in Elderly Patients: Comparison LENOXe™ (xénon 100% v/v) Versus SEVOFLURANE
Brief Title: Hemodynamic Stability During Carotid Endarterectomy.Comparison of LENOXe™ (Xenon 100% v/v) Versus Sevoflurane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALS-8-09-A-401; EUDRACT 2009-012810-29
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hemodynamic Stability
Keywords: hemodynamic stability; xenon; carotid surgery; general anesthesia
MeSH Terms: interventions — Xenon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sévoflurane (Active Comparator): hypnotic use in standard general anesthesia
  Interventions: Drug: sévoflurane
- LENOXe™ (xénon 100 % v/v) (Experimental): Safety of use in terms of hemodynamic stability to the LENOXe™ (xénon 100 % v/v) within the framework of the carotid surgery on the old person
  Interventions: Drug: xenon

INTERVENTIONS:
Drug: xenon — Inhalational gas; dose allowed: 60 % Xenon; the duration of the treatment will be defined through anesthesia-time for a carotid surgery
  Arms: LENOXe™ (xénon 100 % v/v)
Drug: sévoflurane — Inhalation gas; dose allowed: 1,4 %; the duration of the treatment will be defined through anesthesia-time for a carotid surgery
  Arms: sévoflurane

SUMMARY:
The purpose of this study is to compare the hemodynamics effects of two usual hypnotic agents (LENOXe ™ (xenon 100 % v/v) and sevoflurane) during a general anesthesia for carotid endarterectomy in elderly patients. The hypothesis is that the use of the LENOXe ™ (xenon 100 % v/v) allows to obtain per-operating hemodynamic stability non inferior than with sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 55 years, status ASA II
* Carotid endarterectomy elected surgery
* Signed informed consent

Exclusion Criteria:

Related to the patients:

* Histories of hypersensibility in both products used in the study
* uncontrolled arterial High Blood Pressure in the preoperative anaesthesia screening
* Severe cardiac failure (FEVG < 30 %)
* Major lung or airways disease and\or required per-operating FiO2> 35 %
* Elevated intracranial pressure
* Pregnancy, breast feeding
* Major protected, under supervision, under guardianship
* Every patient entering within the framework of the contraindications indicated to §4.3 of the summary of the characteristics of tested products (LENOXe ™ (xenon 100 % v/v), sevoflurane)

Related to the surgery:

* Controlateral carotid stenosis superior to 70 % and\or preoperative indication in the implementation per-operating of a carotid shunt
* Surgery realized within the framework of an emergency
* Combined Surgery

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Standard deviation of the values of systolic blood pressure (SBP)collected per-operatively every minutes(BIOPAC ® MP150) Values of SBP over or under thresholds during and out of the clamping period, if so vasopressive/ hypotensive treatment used | Pre-op, every min from 1-90 min during maintenance phase

SECONDARY OUTCOMES:
cardiovascular, general, hepatic and renal tolerance to xenon. Quality and time of awakening, recovery index (IR);Post-op pain (EVA)and consumption of analgesic; Inflammatory Syndrome (cytokine profile); Subjective comfort of the patient | During the whole anesthetic procedure and the postoperating time until 24 hours after discharge from the recovery room / intensive care unit and return to the ward

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CORIAT, Pr, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Hospital Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Hemodynamic stability of xenon during general anaesthesia for carotid endariectomia in old patientsJune 2011European Journal of Anaesthesiology 28:45DOI:10.1097/00003643-201106001-00138 Yannick Le Manach, G. DouffléJ. P. Goarin, Irene Santos Cristina